CLINICAL TRIAL: NCT06899204
Title: A Prospective, Multi-center Observational Study Characterizing Clinical Outcomes of Patients Receiving Abrocitinib for Moderate-to-severe Atopic Dermatitis Who Had an Inadequate Response (or Intolerance) to ≤2 Previous Biologic Therapies Approved for Moderate-to-severe Atopic Dermatitis
Brief Title: Real World Efficiency of Abrocitinib Treatment at Patients With Moderate to Severe Atopic Dermatitis Who Had Inadequate Response to Previous Biologic Therapies.
Status: Not yet recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451125; JADE-ADVANCED (Other: Alias Study Number)
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis, Unspecified; Dermatitis, Atopic
Keywords: Real world efficacy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — abrocitinib

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Patients that are taking treatment with abrocitinib for moderate to severe atopic dermatitis.
  Interventions: Drug: Abrocitinib

INTERVENTIONS:
Drug: Abrocitinib — Study Drug for Observational Data Collection.
  Other Names: Cibinqo

SUMMARY:
This is a prospective, multi-center observational study characterizing clinical and patient reported outcomes of patients receiving abrocitinib for moderate-to-severe atopic dermatitis (M2S AD) who had inadequate response (or intolerance) to ≤2 previous biologic therapies approved for M2S AD in the United States.

The aim of this study is to measure the effectiveness of abrocitinib in a real-world setting in patients with moderate-to-severe atopic dermatitis, with inadequate response or intolerance to ≤2 biologic therapies.

ELIGIBILITY:
This NI study will enroll 150 patients from approximately 15 sites across the US. The study population eligible for enrollment includes adult and adolescent patients aged ≥12 years diagnosed with moderate to severe AD who receive at least one dose of abrocitinib and satisfy the inclusion and exclusion criteria. Patients who had inadequate response or intolerance to previous ≤2 biologic therapies will be included in this study as there is a lack of effectiveness data for abrocitinib in these patients. As this will be an observational study, there will be no sampling and all patients that meet the inclusion and exclusion criteria will be recruited consequently. The study will be open for enrollment for approximately 12 months after the first patient has been enrolled. Regarding the inclusion and exclusion criteria, in the real-world setting recruitment may be slower than expected, thus depending on the observed enrollment rate, the enrollment period and number of sites may be reassessed and revised during the study.

9.2.1. Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Participants who have chronic AD that has been present for ≥1 year before screening.
2. Male and female patients aged >12 years at baseline.
3. Patients with diagnosis of moderate-to-severe atopic dermatitis confirmed by a certified dermatologist, who are prescribed abrocitinib for use in accordance with the product label (USPI) and independently of the decision to enroll the patient in this study
4. Patients who have inadequate responses or are intolerant to ≤2 previous biologic therapy approved for M2S AD. (Patients shall have had an inadequate response and/or intolerance to at least one, but no more than 2 biologic therapies approved for moderate-to-severe AD)
5. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study. Following receipt of oral and written information about the study, the adolescent (depending on local institutional review board/independent ethics committee requirements) must provide assent, and one or both (according to local regulations) parents or guardians of the child must provide signed informed consent before any study-related activity is carried out.
6. Patients, who in the opinion of the investigator, are willing and able to comply with regular clinic visits as per standard practice at the site and agree to complete PRO questionnaires and other patient completed questions.

9.2.2. Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

1. Patients, that currently have active forms of other inflammatory skin diseases, other than AD or have evidence of skin conditions (eg, psoriasis, seborrheic dermatitis, Lupus) at the time of Day 1 that would interfere with evaluation of atopic dermatitis or response to treatment.
2. Patients previously treated with abrocitinib or other oral/systemic JAK inhibitors
3. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family.
4. Patient eligibility should be reviewed, documented, and confirmed by an appropriately qualified member of the investigator's study team before patients are enrolled in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population eligible for enrollment includes adult and adolescent patients aged ≥12 years diagnosed with moderate to severe AD who receive at least one dose of abrocitinib.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving EASI-75 improvement from baseline at Week 16 after index date | Baseline, week 16
  EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each 4 body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD
Percentage of patients achieving ≥ 4-point improvement in Peak Pruritus Numerical Rating Scale (PP-NRS) collected daily all through the study from baseline at Week 2 by e-diary assessment | Baseline, week 2
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.

SECONDARY OUTCOMES:
Percentage of patients achieving EASI-75, 90 and 100 from baseline at Week 4 and 16 after index date | Baseline, week 4, week 16
  EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each 4 body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD
Percentage of patients achieving v-IGA response of Clear (0) or Almost Clear (1) and ≥ 2 points improvement from baseline at Week 4 and 16 after index date | Baseline, week 4, week 16
  Validated IGA assesses severity of participant's AD on a 5 point scale. 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting and 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Higher scores indicating more severity of AD. Assessment excluded soles, palms and scalp.
Change from baseline in total percentage of BSA at week 4 and 16 | Baseline, week 4, week 16
  4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%, with higher values representing greater severity of AD
Percentage of patients achieving Peak Pruritus Numerical Rating Scale (PP-NRS) of 0 or 1 collected daily all through the study at Wk 4, 12 and 16 | Baseline, week 4, 12 and 16
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Percentage of patients achieving PP-NRS-4 at week 2, 4, 12 and 16 from baseline. | Baseline, week 2, 4, 12 and 16
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch
Absolute change from baseline in PP-NRS score at week 2 | Baseline, week2
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch
Proportion of patients overall "Very Satisfied" and "Satisfied" with abrocitinib at Wk 4, 12 and 16 with TSQM-9 | Baseline, week 4, 12 and 16
  TSQM-9 is a generic satisfaction assessment instrument to measure patient satisfaction with the medication taken.
Percentage of patients that report symptoms to be "minimal" or "absent" on the patient global impression of severity at week 4, 12 and 16 | Baseline week 4, 12 and 16
  PGI-S: A single-item PRO questionnaire assessing overall current disease severity on a 7-point verbal response scale
Change from baseline in Medical Outcomes Study - Sleep Scale (MOS-Sleep Scale) at Wk 4, 12 and 16 | Baseline, week 4, 12 and 16
  The MOS Sleep Scale is a 12-item measure that is segregated into subscales addressing seven sleep domains (i.e. sleep disturbance, snoring, short of breath or headache, adequacy of sleep, somnolence, sleep problems index I and sleep problems index II). An additional single item assessed quantity of sleep. Each of the sleep domains were scored on a range of 0 to 100, and higher scores indicated worse outcomes. The quantity of sleep scores ranged from 0 to 24 (number of hours slept). Change from baseline scores for each individual sleep domain and quantity of sleep are reported in this outcome measure.
Percentage of Participants with an ADCT Total Score Reduction ≥ 5 from baseline at week 4, 12 and 16 | Baseline, week 4, 12 and 16
  The ADCT is a validated, brief and easily scored tool for use in clinical practice and clinical research to evaluate 6 symptoms and effects associated with AD over the past week.
Percentage of Participants Achieving Improvement (reduction) in DLQI/CDLQI of ≥ 4 points vs baseline at week 4, 12 and 16 | Baseline week 4, 12 and 16
  CDLQI is a 10-item questionnaire that measures the impact of skin disease on adolescents (aged 12-17 years) quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. CDLQI total score was the sum of individual scores of question 1-10 and ranges from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of children. DLQI is the adult version of the same index.
Observational change in pigment alteration from baseline at week 4 and 16 by visual assessment of available photography | Baseline, week 4, and 16
  Physician visual evaluation of the pigmentation changes of the AD lesions.
Cilinical Characteristics: Type of prior AD treatment at specific medication level and Route of Administration | Baseline
Demographic charasteristics: Number/percentage of patients by age, sex, race, ethnicity, socioeconomic status, state of residence | Baseline
Clinical Characteristics: Number/percentage of patients by smoking status, medical history | Baseline
Clinical Characteristics: Duration of prior therapy/frequency | Baseline
Clinical Characteristics: Total number of AD treatments used prior to abrocitinib initiation | Baseline
Clinical characteristics : Reason for switching to abrocitinib from previous biologic | Baseline
Outcome: Assessment of efficacy in patients who received a dose change after baseline visit (dose increase or decrease) | Week 4, week 16
Assess early improvement in itch (within min/hrs) after first dose | Baseline, day 1 after index date
  Patients will be asked when they realized improvement in their itch within the first day of abrocitinib treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.